CLINICAL TRIAL: NCT02043106
Title: Plantar Cutaneous Stimulation Used to Elicit Muscle Activity in Individuals With Incomplete Spinal Cord Injury
Brief Title: Can Vibration Stimulation of the Foot Sole Activate Leg Muscles?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Dr. Stephen Perry, Assoicate Professor, Wilfrid Laurier University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC_SCIPS
Record Dates: First submitted 2013-11-25; First posted 2014-01-23 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- spinal cord injury (Experimental): Individuals who have sustained an incomplete spinal cord injury
  Interventions: Other: plantar vibration
- non-spinal cord injury (Active Comparator): Individuals who have not sustained a spinal cord injury
  Interventions: Other: plantar vibration

INTERVENTIONS:
Other: plantar vibration

SUMMARY:
Participants will be asked to complete three different tests (standing, stepping and assisted walking) and will experience three different experimental conditions during each test. The three conditions are types of vibratory plantar cutaneous stimulation, which include no vibratory stimulation, submaximal vibratory stimulation and supramaximal vibratory stimulation. In the first condition, participants will experience no stimulation applied to any part of the body. In the second condition, a submaximal vibratory stimulus will be delivered at 90% of the participant's threshold to the surface of the foot. In the third condition, a supramaximal vibratory stimulus will be delivered at three times the participant's threshold. The hypothesis is that this plantar stimulation (90% threshold and supramaximal) will elicit increased muscle activity during these tests. If the hypothesis is positive then this protocol will also be presented in incomplete spinal cord injuried participants.

ELIGIBILITY:
Inclusion Criteria:

* no spinal cord injury

Exclusion Criteria:

* any musculoskeletal or neurological disease that affects movement or balance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Muscle activity | up to 2 months after experiment
  Muscle activity will be measured by electromyography equipment (two electrodes placed on the muscle belly) and then the outcome measures will be the description of both the timing (relative to task onset) and magintude of muscle activity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Perry, PhD, Study Director — Wilfrid Laurier University
Locations (1):
- Biomechanics Lab, Wilfrid Laurier University, Waterloo, Ontario, Canada